CLINICAL TRIAL: NCT00711529
Title: Comparison of Hypnotherapy Versus Gabapentin in the Treatment of Hot Flashes in Breast Cancer Survivors or Women at Risk of Developing Breast Cancer.
Brief Title: Pilot Study Comparing Hypnotherapy and Gabapentin for Hot Flashes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Shannon MacLaughlan, Shannon MacLaughlan, M.D., Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 08-0057
Record Dates: First submitted 2008-07-03; First posted 2008-07-09 (Estimated); Results first posted 2013-06-24 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-05

CONDITIONS: Breast Cancer; Hot Flashes
Keywords: hot flashes; breast cancer; Hypnotherapy; Quality of Life; Gabapentin
MeSH Terms: conditions — Breast Neoplasms; Hot Flashes | interventions — Hypnosis; Mind-Body Therapies; Gabapentin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypnotherapy (Experimental): Patients randomized to the experimental arm were scheduled for three one-hour inductions by a single hypnotherapist, each one week apart. Standardized outlines were used for each induction. The second and third sessions also began with a standardized induction, followed by the establishment of an "anchor," or physical reference point (forefinger to thumb), used to invoke images of coolness, which were individualized according to patient preference.
  Patients were also instructed by the same hypnotherapist in self-hypnosis and guided imagery techniques to be used at home with the assistance of standardized audio compact disks. Participation lasted eight weeks.
  Interventions: Behavioral: Hypnotherapy
- Gabapentin (Active Comparator): Patients randomized to the gabapentin arm were prescribed 900mg of the drug daily (300 mg by mouth three times daily).
  Interventions: Drug: gabapentin

INTERVENTIONS:
Behavioral: Hypnotherapy — Patients randomized to the hypnosis arm of the study will undergo individually three one-hour sessions with a certified hypnotherapist. These sessions will be one week apart. surveys. The therapist will be prohibited from asking subjects about clinical responses to the hypnosis sessions. The patients will also be instructed on self-hypnosis techniques to be used at home.
  Other Names: hypnosis; mind-body therapy
  Arms: Hypnotherapy
Drug: gabapentin — Patients randomized to the gabapentin arm will be prescribed 900mg of the drug daily (300 mg by mouth three times daily). This dose has been shown to be more effective than 300mg daily. Larger doses have not been evaluated in this population, and may be associated with a more significant side-effect profile. The prescription for gabapentin will be provided at the patient's enrollment appointment. The patients will take gabapentin as prescribed daily for the study-enrollment period, which is 8 weeks.
  Other Names: Neurontin; gabarone
  Arms: Gabapentin

SUMMARY:
Premenopausal women with breast cancer who receive endocrine therapy (e.g. tamoxifen) and/or chemotherapy are at risk for experiencing premature menopause because of their treatment. The resulting symptoms, most notably hot flashes, can cause significant detriment to a patient's quality of life. Treatment for menopausal symptoms with the gold standard of hormone replacement therapy is not done routinely as it is unclear whether it can increase risk of tumor recurrence. In addition, many medical oncologists feel it is contraindicated in this population, especially among women whose breast cancers have estrogen receptors. This has lead to an increased interest in options other than estrogen replacement in the treatment of hot flashes, though most investigations of alternative medications have shown a suboptimal response.

Recent studies have suggested that non-drug treatments using alternative or complementary therapies may be effective. Specifically, hypnosis has been promoted as a means to control hot flashes, though it has not been tested in a randomized fashion. In accordance with the National Cancer Institute's recent initiatives to expand the goals of clinical trials to include symptom management studies, our purpose is to evaluate the role of complementary and alternative therapies for improvement of symptoms in women with breast cancer. Specifically, we plan to evaluate the use of hypnotherapy for the treatment of therapy-induced hot flashes in breast cancer survivors. We intend to recruit 60 women into a pilot feasibility trial comparing hypnotherapy to the drug gabapentin (Neurontin®) for the treatment of therapy-induced hot flashes in eligible women who are receiving care at the Breast Health Center. We have chosen gabapentin based on recent studies showing it may be an effective non-estrogen treatment for this indication.

We will identify patients who are experiencing at least one daily hot flash as a result of the treatment they received for their breast cancer for participation. When enrolled, they will be randomized into either the treatment arm, in which they will receive daily gabapentin, or the experimental arm, in which they will undergo weekly hypnotherapy.

Our study hypothesis is that hypnotherapy will be more effective than gabapentin in the control of hot flashes in this population.

DETAILED DESCRIPTION:
Roughly half of women diagnosed with pre-menopausal breast cancer will have hormone receptor-positive tumors, which will make them candidates for anti-estrogen therapies. Both endocrine therapy and ovarian ablation have also been shown to improve outcomes in this population.

Hot flashes are a frequent side effect in women receiving anti-estrogen therapy for breast cancer, and have been shown to have a significant impact on patients' quality of life. For example, it has been reported that hot flashes in breast cancer survivors are more severe and result in a more significant impact on quality of life measures when compared with healthy women.

Hormone replacement, the gold standard for the treatment of hot flashes in postmenopausal women, is contraindicated in this population. Non-hormonal drug therapies have been explored for the treatment of hot flashes in this population of women with moderate results. In randomized controlled trials, venlafaxine has been shown to reduce self-reported hot flashes in patients with breast cancer by 25-61%. However, selective serotonin re-uptake inhibitors (SSRIs) and selective norepinephrine re-uptake inhibitors (SNRIs) may interfere with the metabolism of tamoxifen, a common treatment for estrogen-receptor positive breast cancers, by inhibiting the cytochrome P450 2D6 (CYP2D6) enzyme. Gabapentin is a gamma-aminobutyric acid (GABA) analogue commonly used for the treatment of seizure disorders and neuropathic pain. There is some evidence to demonstrate its efficacy in hot flashes to be equivalent to estrogen and superior to antidepressants in postmenopausal women.

In a pilot study of 22 women with breast cancer on tamoxifen, the use of gabapentin for four weeks reduced the frequency of hot flashes by 44.2%, and decreased the hot flash severity scores by 52.6%. These results were confirmed in a larger study of 420 breast cancer survivors who were randomized to receive gabapentin 300mg/d, gabapentin 900mg/d, or placebo. The 900mg/d dose of gabapentin was the most effective; decreasing the frequency of hot flashes by 49% at four weeks. In the group receiving 900mg of gabapentin daily, there was a 12% withdrawal rate at 4 weeks, and 17% at 8 weeks, owing to side effects and subjective inefficacy.

Hypnosis or hypnotherapy, defined as the induction of a deeply relaxed condition that allows the patient to suspend critical faculties and allow suggestibility, has been shown to be effective in not only reducing the daily frequency of hot flashes (by 59%), but also in improving quality of life variables such as insomnia in patients with breast cancer. However, this therapy has never been compared directly to pharmacotherapy in the treatment of therapy-induced hot flashes in patients with breast cancer.

In response to the NCI's 2006 initiatives to expand the goals of clinical trials and include symptom management studies, we are interested in evaluating the role of complementary and alternative therapies for improvement of symptoms in women with breast cancer. This trial is to determine whether hypnotherapy, administered in a standard way, can improve the frequency of hot flashes and breast cancer specific quality of life in women diagnosed with pre-menopausal breast cancer. We propose to evaluate this through a pilot feasibility study which will randomize participants to an eight week course of gabapentin or hypnosis.

ELIGIBILITY:
Inclusion criteria:

* Women with histologic confirmation of a diagnosis of infiltrating carcinoma of the breast are eligible for participation.
* Women with non-invasive or pre-invasive lesions of the breast, including but not limited to ductal carcinoma in situ (DCIS), atypical ductal hyperplasia (ADH) or lobular carcinoma in situ (LCIS) are eligible for participation.
* Women with a known breast cancer susceptibility gene (eg, BRCA) mutation or strong family history of breast cancer are eligible.
* Any woman age 60 years or more who cannot take estrogen therapy because of a real or perceived risk of developing breast cancer are eligible.
* Women under the age of 60 with a Gail model score of 1.6% or more are eligible.
* Subjective report of at least one daily hot flash.
* Able to provide voluntary informed consent.
* ≥ 18 years-old. There will be no upper limit for age inclusion.
* Karnofsky performance status > 70%.
* Women with a history of breast cancer must have undergone treatment with curative intent.
* ≥ 4 weeks from completion of chemotherapy or radiation therapy, where appropriate.
* adequate hematopoietic function (ANC ≥ 1500/mm3; Platelets ≥ 100,000/mm3; Hemoglobin ≥ 8 g/dL)
* adequate renal and hepatic function [Bilirubin ≤ 1.5 times upper limit of normal (ULN), serum glutamic-oxaloacetic transaminase (SGOT) ≤ 2.5x ULN, Alkaline phosphatase ≤ 2.5x ULN, and Creatinine ≤ 2x ULN].
* No clinical evidence of disease (complete remission).
* Patients receiving neoadjuvant therapy will be eligible following completion of all adjuvant chemotherapy if indicated.
* Patients receiving hormonal therapy in lieu of or following chemotherapy will be eligible to participate.
* Patients must have access to a compact disk player.

Exclusion criteria:

* History or active secondary cancer within the last 5 years (except for superficial basal cell skin cancers).
* Any residual chemotherapy-induced CTCv3.0 Grade 2 or greater non-hematological toxicity.
* Unable to give informed consent or unable to adhere to protocol.
* Any serious medical or psychiatric illness likely to interfere with participation in this clinical study, concurrent uncontrolled illness, or ongoing or active infection will be excluded.
* Any history of alcohol or drug abuse.
* Allergy to gabapentin.
* History of seizure disorder.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon D MacLaughlan, MD, Principal Investigator — Women & Infants' Hospital of Rhode Island; Don S Dizon, MD, Principal Investigator — Women & Infants' Hospital of Rhode Island
Locations (1):
- Breast Health Center, Program in Women's Oncology, Women & Infants' Hospital of Rhode Island, Providence, Rhode Island, United States

REFERENCES:
- [Background] Goldhirsch A, Gelber RD, Castiglione M. The magnitude of endocrine effects of adjuvant chemotherapy for premenopausal breast cancer patients. The International Breast Cancer Study Group. Ann Oncol. 1990;1(3):183-8. doi: 10.1093/oxfordjournals.annonc.a057718. PMID 2261364
- [Background] Anderson WF, Jatoi I, Devesa SS. Distinct breast cancer incidence and prognostic patterns in the NCI's SEER program: suggesting a possible link between etiology and outcome. Breast Cancer Res Treat. 2005 Mar;90(2):127-37. doi: 10.1007/s10549-004-3777-3. PMID 15803359
- [Background] Bines J, Oleske DM, Cobleigh MA. Ovarian function in premenopausal women treated with adjuvant chemotherapy for breast cancer. J Clin Oncol. 1996 May;14(5):1718-29. doi: 10.1200/JCO.1996.14.5.1718. PMID 8622093
- [Background] Del Mastro L, Venturini M, Sertoli MR, Rosso R. Amenorrhea induced by adjuvant chemotherapy in early breast cancer patients: prognostic role and clinical implications. Breast Cancer Res Treat. 1997 Apr;43(2):183-90. doi: 10.1023/a:1005792830054. PMID 9131274
- [Background] Couzi RJ, Helzlsouer KJ, Fetting JH. Prevalence of menopausal symptoms among women with a history of breast cancer and attitudes toward estrogen replacement therapy. J Clin Oncol. 1995 Nov;13(11):2737-44. doi: 10.1200/JCO.1995.13.11.2737. PMID 7595732
- [Background] Jonat W, Kaufmann M, Sauerbrei W, Blamey R, Cuzick J, Namer M, Fogelman I, de Haes JC, de Matteis A, Stewart A, Eiermann W, Szakolczai I, Palmer M, Schumacher M, Geberth M, Lisboa B; Zoladex Early Breast Cancer Research Association Study. Goserelin versus cyclophosphamide, methotrexate, and fluorouracil as adjuvant therapy in premenopausal patients with node-positive breast cancer: The Zoladex Early Breast Cancer Research Association Study. J Clin Oncol. 2002 Dec 15;20(24):4628-35. doi: 10.1200/JCO.2002.05.042. PMID 12488406
- [Background] International Breast Cancer Study Group (IBCSG); Castiglione-Gertsch M, O'Neill A, Price KN, Goldhirsch A, Coates AS, Colleoni M, Nasi ML, Bonetti M, Gelber RD. Adjuvant chemotherapy followed by goserelin versus either modality alone for premenopausal lymph node-negative breast cancer: a randomized trial. J Natl Cancer Inst. 2003 Dec 17;95(24):1833-46. doi: 10.1093/jnci/djg119. PMID 14679153
- [Background] Northouse LL. Breast cancer in younger women: effects on interpersonal and family relations. J Natl Cancer Inst Monogr. 1994;(16):183-90. PMID 7999463
- [Background] Ganz PA, Rowland JH, Desmond K, Meyerowitz BE, Wyatt GE. Life after breast cancer: understanding women's health-related quality of life and sexual functioning. J Clin Oncol. 1998 Feb;16(2):501-14. doi: 10.1200/JCO.1998.16.2.501. PMID 9469334
- [Background] Ganz PA, Greendale GA, Petersen L, Kahn B, Bower JE. Breast cancer in younger women: reproductive and late health effects of treatment. J Clin Oncol. 2003 Nov 15;21(22):4184-93. doi: 10.1200/JCO.2003.04.196. PMID 14615446
- [Background] Avis NE, Crawford S, Manuel J. Quality of life among younger women with breast cancer. J Clin Oncol. 2005 May 20;23(15):3322-30. doi: 10.1200/JCO.2005.05.130. PMID 15908646
- [Background] Carpenter JS, Andrykowski MA, Cordova M, Cunningham L, Studts J, McGrath P, Kenady D, Sloan D, Munn R. Hot flashes in postmenopausal women treated for breast carcinoma: prevalence, severity, correlates, management, and relation to quality of life. Cancer. 1998 May 1;82(9):1682-91. PMID 9576289
- [Background] Loprinzi CL, Kugler JW, Sloan JA, Mailliard JA, LaVasseur BI, Barton DL, Novotny PJ, Dakhil SR, Rodger K, Rummans TA, Christensen BJ. Venlafaxine in management of hot flashes in survivors of breast cancer: a randomised controlled trial. Lancet. 2000 Dec 16;356(9247):2059-63. doi: 10.1016/S0140-6736(00)03403-6. PMID 11145492
- [Background] Carpenter JS, Storniolo AM, Johns S, Monahan PO, Azzouz F, Elam JL, Johnson CS, Shelton RC. Randomized, double-blind, placebo-controlled crossover trials of venlafaxine for hot flashes after breast cancer. Oncologist. 2007 Jan;12(1):124-35. doi: 10.1634/theoncologist.12-1-124. PMID 17227907
- [Background] Jin Y, Desta Z, Stearns V, Ward B, Ho H, Lee KH, Skaar T, Storniolo AM, Li L, Araba A, Blanchard R, Nguyen A, Ullmer L, Hayden J, Lemler S, Weinshilboum RM, Rae JM, Hayes DF, Flockhart DA. CYP2D6 genotype, antidepressant use, and tamoxifen metabolism during adjuvant breast cancer treatment. J Natl Cancer Inst. 2005 Jan 5;97(1):30-9. doi: 10.1093/jnci/dji005. PMID 15632378
- [Background] Reddy SY, Warner H, Guttuso T Jr, Messing S, DiGrazio W, Thornburg L, Guzick DS. Gabapentin, estrogen, and placebo for treating hot flushes: a randomized controlled trial. Obstet Gynecol. 2006 Jul;108(1):41-8. doi: 10.1097/01.AOG.0000222383.43913.ed. PMID 16816054
- [Background] Loprinzi CL, Kugler JW, Barton DL, Dueck AC, Tschetter LK, Nelimark RA, Balcueva EP, Burger KN, Novotny PJ, Carlson MD, Duane SF, Corso SW, Johnson DB, Jaslowski AJ. Phase III trial of gabapentin alone or in conjunction with an antidepressant in the management of hot flashes in women who have inadequate control with an antidepressant alone: NCCTG N03C5. J Clin Oncol. 2007 Jan 20;25(3):308-12. doi: 10.1200/JCO.2006.07.5390. Epub 2006 Dec 4. PMID 17146104
- [Background] Pandya KJ, Thummala AR, Griggs JJ, Rosenblatt JD, Sahasrabudhe DM, Guttuso TJ, Morrow GR, Roscoe JA. Pilot study using gabapentin for tamoxifen-induced hot flashes in women with breast cancer. Breast Cancer Res Treat. 2004 Jan;83(1):87-9. doi: 10.1023/B:BREA.0000010676.54597.22. PMID 14997058
- [Background] Pandya KJ, Morrow GR, Roscoe JA, Zhao H, Hickok JT, Pajon E, Sweeney TJ, Banerjee TK, Flynn PJ. Gabapentin for hot flashes in 420 women with breast cancer: a randomised double-blind placebo-controlled trial. Lancet. 2005 Sep 3-9;366(9488):818-24. doi: 10.1016/S0140-6736(05)67215-7. PMID 16139656
- [Background] Elkins G, Marcus J, Stearns V, Hasan Rajab M. Pilot evaluation of hypnosis for the treatment of hot flashes in breast cancer survivors. Psychooncology. 2007 May;16(5):487-92. doi: 10.1002/pon.1096. PMID 17048223
- [Background] Elkins G, Marcus J, Palamara L, Stearns V. Can hypnosis reduce hot flashes in breast cancer survivors? A literature review. Am J Clin Hypn. 2004 Jul;47(1):29-42. doi: 10.1080/00029157.2004.10401473. PMID 15376607
- [Background] Younus J, Simpson I, Collins A, Wang X. Mind control of menopause. Womens Health Issues. 2003 Mar-Apr;13(2):74-8. doi: 10.1016/s1049-3867(02)00196-2. PMID 12732444
- [Background] Buettner C, Kroenke CH, Phillips RS, Davis RB, Eisenberg DM, Holmes MD. Correlates of use of different types of complementary and alternative medicine by breast cancer survivors in the nurses' health study. Breast Cancer Res Treat. 2006 Nov;100(2):219-27. doi: 10.1007/s10549-006-9239-3. Epub 2006 Jul 5. PMID 16821087
- [Background] Daut RL, Cleeland CS, Flanery RC. Development of the Wisconsin Brief Pain Questionnaire to assess pain in cancer and other diseases. Pain. 1983 Oct;17(2):197-210. doi: 10.1016/0304-3959(83)90143-4. PMID 6646795
- [Background] Hann DM, Jacobsen PB, Azzarello LM, Martin SC, Curran SL, Fields KK, Greenberg H, Lyman G. Measurement of fatigue in cancer patients: development and validation of the Fatigue Symptom Inventory. Qual Life Res. 1998 May;7(4):301-10. doi: 10.1023/a:1024929829627. PMID 9610214
- [Background] Carpenter JS. The Hot Flash Related Daily Interference Scale: a tool for assessing the impact of hot flashes on quality of life following breast cancer. J Pain Symptom Manage. 2001 Dec;22(6):979-89. doi: 10.1016/s0885-3924(01)00353-0. PMID 11738160
- [Background] Groenvold M, Klee MC, Sprangers MA, Aaronson NK. Validation of the EORTC QLQ-C30 quality of life questionnaire through combined qualitative and quantitative assessment of patient-observer agreement. J Clin Epidemiol. 1997 Apr;50(4):441-50. doi: 10.1016/s0895-4356(96)00428-3. PMID 9179103
- [Background] Osoba D, Rodrigues G, Myles J, Zee B, Pater J. Interpreting the significance of changes in health-related quality-of-life scores. J Clin Oncol. 1998 Jan;16(1):139-44. doi: 10.1200/JCO.1998.16.1.139. PMID 9440735
- [Background] Sprangers MA, Groenvold M, Arraras JI, Franklin J, te Velde A, Muller M, Franzini L, Williams A, de Haes HC, Hopwood P, Cull A, Aaronson NK. The European Organization for Research and Treatment of Cancer breast cancer-specific quality-of-life questionnaire module: first results from a three-country field study. J Clin Oncol. 1996 Oct;14(10):2756-68. doi: 10.1200/JCO.1996.14.10.2756. PMID 8874337
- [Background] Hedeker D, Mermelstein RJ. Application of random-effects regression models in relapse research. Addiction. 1996 Dec;91 Suppl:S211-29. PMID 8997794
- [Background] Hedeker D, Gibbons RD. MIXREG: a computer program for mixed-effects regression analysis with autocorrelated errors. Comput Methods Programs Biomed. 1996 May;49(3):229-52. doi: 10.1016/0169-2607(96)01723-3. PMID 8800609
- [Background] Sloan JA, Loprinzi CL, Novotny PJ, Barton DL, Lavasseur BI, Windschitl H. Methodologic lessons learned from hot flash studies. J Clin Oncol. 2001 Dec 1;19(23):4280-90. doi: 10.1200/JCO.2001.19.23.4280. PMID 11731510
- [Derived] Maclaughlan David S, Salzillo S, Bowe P, Scuncio S, Malit B, Raker C, Gass JS, Granai CO, Dizon DS. Randomised controlled trial comparing hypnotherapy versus gabapentin for the treatment of hot flashes in breast cancer survivors: a pilot study. BMJ Open. 2013 Sep 10;3(9):e003138. doi: 10.1136/bmjopen-2013-003138. PMID 24022390

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between September 2008 and September 2010, 73 women were screened for this study. Fourteen women were deemed ineligible and 32 decided not to participate. A total of 27 women were randomized to receive treatment, 14 to gabapentin and 13 to hypnotherapy.
Groups:
- Hypnotherapy: Patients randomized to the hypnosis arm of the study will undergo individually three one-hour sessions with a certified hypnotherapist. These sessions will be one week apart. Patients will also be instructed on the use of self-hypnosis techniques to use at home.
- Gabapentin: Patients randomized to the gabapentin arm will be prescribed 900mg of the drug daily (300 mg by mouth three times daily).
Period: Overall Study
Arm/Group | Hypnotherapy | Gabapentin
Started | 13 | 14
Completed | 9 (2 women lost their hot flash diary, so only 7 patients were evaluable for primary endpoint.) | 8
Not Completed | 4 | 6
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 6

BASELINE CHARACTERISTICS:
Population: Of the 13 women randomized to the hypnotherapy arm, 2 women were ineligible and therefore not included in analysis. Two women were unable to initate treatment and did not submit diaries. Two women lost their diaries, leaving 7 diaries for analysis. Of the 14 women randomized to receive gabapentin, 6 dropped out and did not submit diaries.
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypnotherapy | Gabapentin | Total
Number analyzed (Participants) | 11 | 14 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 14 | 25
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 14 | 25
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Daily Hot Flashes
Description: Patients kept daily diaries of their hot flashes. The absolute number of hot flashes in a 24 hour period is "number of daily hot flashes." The median number was calculated for each week of data. The median number of daily hot flashes for the first week (7 days) of participation is used as baseline. The median number of daily hot flashes for the fourth week (over 7 day interval) is reported for the week four time point. The median number of daily hot flashes for the eighth week (over 7 day interval) is reported for the week eight time point (study completion). Of the 13 women randomized to the hypnotherapy arm, 2 women were ineligible and therefore not included in analysis. Two women were unable to initiate treatment and did not submit diaries. An additional two women completed treatment but lost their diaries, leaving 7 diaries for analysis at baseline. Of the 14 randomized to receive gabapentin, 6 dropped out of the study and did not submit diaries.
Time Frame: Baseline
Measure: Median (Full Range); unit: daily hot flashes
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 7 | 8
daily hot flashes | 5 [2 to 11] | 4.5 [2 to 9]

2. Primary Outcome: Number of Daily Hot Flashes
Description: Patients kept daily diaries of their hot flashes. The absolute number of hot flashes in a 24 hour period is "number of daily hot flashes." The median number was calculated for each week of data. The median number of daily hot flashes for the first week (7 days) of participation is used as baseline. The median number of daily hot flashes for the fourth week (over 7 day interval) is reported for the week four time point. The median number of daily hot flashes for the eighth week (over 7 day interval) is reported for the week eight time point (study completion). A total of 15 diaries were submitted (7 hypnotherapy, 8 gabapentin). One person in each arm stopped recording in her diary before the 4 week mark.
Time Frame: Week 4
Measure: Median (Full Range); unit: daily hot flashes
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 6 | 7
daily hot flashes | 4 [1 to 7] | 4 [2 to 9]

3. Primary Outcome: Number of Daily Hot Flashes
Description: Patients kept daily diaries of their hot flashes. The absolute number of hot flashes in a 24 hour period is "number of daily hot flashes." The median number was calculated for each week of data. The median number of daily hot flashes for the first week (7 days) of participation is used as baseline. The median number of daily hot flashes for the fourth week (over 7 day interval) is reported for the week four time point. The median number of daily hot flashes for the eighth week (over 7 day interval) is reported for the week eight time point (study completion). One woman in the hypnotherapy arm and 3 women in the gabapentin arm stopped keeping their diary before the 8 week mark.
Time Frame: Week 8
Measure: Median (Full Range); unit: daily hot flashes
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 6 | 5
daily hot flashes | 1 [0 to 7] | 3 [3 to 5.5]

4. Primary Outcome: Hot Flash Severity Score
Description: The patients kept daily hot flash diaries, including the total number of hot flashes they characterized as mild, moderate,severe and very severe. Hot flash severity scores were calculated by assigning one point to each mild hot flash, two points for each moderate hot flash, three points for each severe hot flash and four points for each very severe hot flash. The hot flash severity score for a 24 hour period was the sum of these scores. The score was calculated for each day in the diary. For each subject, median scores were calculated for each week (7 day period) of participation. The median hot flash severity score for the first week was considered the baseline. The median hot flash severity score for the fourth week is considered the week 4 time point. The median hot flash severity score for the eighth week is considered the week 8 time point. The median result for the group was then calculated at each of the timepoints.
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale (severity score)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 7 | 8
units on a scale (severity score) | 10 [2 to 14] | 7.5 [2 to 17.5]

5. Primary Outcome: Hot Flash Severity Score
Description: as for outcome 4
Time Frame: Week 4
Measure: Median (Full Range); unit: units on a scale (severity score)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 6 | 7
units on a scale (severity score) | 6.5 [1 to 11] | 4 [2 to 17.5]

6. Primary Outcome: Hot Flash Severity Score
Description: as for outcome 4
Time Frame: Week 8
Measure: Median (Full Range); unit: units on a scale (severity score)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 6 | 5
units on a scale (severity score) | 1.5 [0 to 12] | 5 [3 to 11.5]

7. Secondary Outcome: Hot Flash Related Daily Interference Score (HFRDIS)
Description: The HFRDIS is a validated survey of 10 questions asking patients to rate ten symptoms on a scale of 0-10. The HFRDIS is a sum of the scores in each category, so that total score can range from 0 (no symptoms) to 100 (10 severe symptoms). These surveys were conducted at the time of enrollment (baseline), after four weeks of treatment, and at the conclusion of the study (8 weeks). All women who were randomized were included in the baseline analysis (with the exception of 2 women excluded from the hypnotherapy arm who were deemed ineligible after randomization).
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale (HFRDIS)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 11 | 14
units on a scale (HFRDIS) | 58 [16 to 64] | 45.5 [11 to 82]

8. Secondary Outcome: Hot Flash Related Daily Interference Score (HFRDIS)
Description: The HFRDIS is a validated survey of 10 questions asking patients to rate ten hot flash-related symptoms on a scale of 0-10. The HFRDIS is a sum of the scores in each category, so that total score can range from 0 (no symptoms) to 100 (10 severe symptoms). These surveys were conducted at the time of enrollment (baseline), after four weeks of treatment, and at the conclusion of the study (8 weeks). Of 11 eligible women in the hypnotherapy arm, 2 never initiated treatment, and 3 did not complete the survey at this time point. Of the 14 eligible women in the gabapentin arm, 3 never initiated treatment, and 3 dropped out of the study before the 4 week time point.
Time Frame: Week 4
Measure: Median (Full Range); unit: units on a scale (HFRDIS)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 6 | 8
units on a scale (HFRDIS) | 25.5 [1 to 57] | 21.5 [0 to 57]

9. Secondary Outcome: Hot Flash Related Daily Interference Score (HFRDIS)
Description: The HFRDIS is a validated survey of 10 questions asking patients to rate ten hot flash-related symptoms on a scale of 0-10. The HFRDIS is a sum of the scores in each category, so that total score can range from 0 (no symptoms) to 100 (10 severe symptoms). These surveys were conducted at the time of enrollment (baseline), after four weeks of treatment, and at the conclusion of the study (8 weeks). All nine women who initiated hypnotherapy treatment completed the survey at the end of 8 weeks. One woman in the gabapentin arm did not submit a survey at 8 weeks.
Time Frame: Week 8
Measure: Median (Full Range); unit: units on a scale (HFRDIS)
Arm/Group | Hypnotherapy | Gabapentin
Number analyzed (Participants) | 9 | 7
units on a scale (HFRDIS) | 26 [0 to 68] | 22 [7 to 41]

ADVERSE EVENTS:
Time Frame: 2 years, 11 months
Arm/Group | Hypnotherapy | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/14
Other Adverse Events (participants affected / at risk) | 0/13 | 0/14

LIMITATIONS AND CAVEATS:
We were unable to meet recruitment goals because of 1) lower-than-anticipated rate of referrals, and 2) subjects' unwillingness to randomization. This resulted in small numbers that limit interpretation of results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No